CLINICAL TRIAL: NCT00374062
Title: Effect of the Subconscious on Mohs Micrographic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Murad Alam, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1253-017
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Mohs Surgery
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Experimental): relaxation tape 1
  Interventions: Behavioral: relaxation therapy 1
- II (Experimental): relaxation tape 2
  Interventions: Behavioral: relaxation therapy 2
- III (Placebo Comparator): relaxation tape 3
  Interventions: Behavioral: relaxation therapy 3

INTERVENTIONS:
Behavioral: relaxation therapy 1 — relaxation therapy 1
  Arms: I
Behavioral: relaxation therapy 2 — relaxation therapy 2
  Arms: II
Behavioral: relaxation therapy 3 — relaxation therapy 3
  Arms: III

SUMMARY:
The goal of this study is to determine if relaxation therapy improves patient satisfaction with Mohs micrographic surgery.

DETAILED DESCRIPTION:
Patients are instructed in relaxation techniques. The goal of this study is to determine how relaxation techniques affect the patient's Mohs micrographic surgery experience.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 and older
* Subjects are undergoing micrographic Mohs surgery for facial basal and squamous cell carcinoma.
* The subjects are in good health.
* The subjects have willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

* Subjects who have wound healing problems.
* Subjects who have had prior Mohs surgery.
* Subjects who are smokers.
* Subjects who are currently using anticoagulation therapy
* Subjects who have a history of bleeding disorders.
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with known mental illness or other psychological conditions, such as psychotic disorders, mood disorders, anxiety disorders, cognitive disorders, depression with psychotic features, dissociative disorders.
* Subjects who are taking medications that may affect healing such as prednisone, or any immunosuppressants.
* Subjects who are immunocompromised.
* Subjects who have Diabetes Mellitus or any other condition determined by the PI to affect healing.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Patient anxiety | 1 day

SECONDARY OUTCOMES:
Scar appearance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Murad Alam, MD, Chicago, Illinois, United States